CLINICAL TRIAL: NCT07247708
Title: Exploring the Correlation Between Workload, Stress Level, and Health Status of Nurses Through Wearable Technology and Shift Data: A Feasibility Study
Brief Title: Mizzou Nurse Workload and Well-Being Study
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Oura Ring (Unknown)
Responsible Party: Principal Investigator, Jennifer Hulett, Associate Professor, University of Missouri-Columbia
Other Study IDs: 2101866; URC-025-19 (Other Grant/Funding Number: University of Missouri Research Council)
Record Dates: First submitted 2025-09-29; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Burnout, Healthcare Workers; Nursing Workload
Keywords: burnout; nursing workload; acute care nursing; physiological stress; job satisfaction; biometric measurement; organizational factors in health care; well-being
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intensive Care Unit: surgical ICU and cardiac ICU RNs
  Interventions: Other: Multimethod data collection
- Medical-Surgical Unit: surgical and cardiovascular units
  Interventions: Other: Multimethod data collection

INTERVENTIONS:
Other: Multimethod data collection — Participants will contribute data through three integrated sources: workload metrics (workforce management software to assess patient acuity and shift characteristics); biometric monitoring (physiological data collected via the Oura Ring); and self-report surveys and semi-structured interviews.
  Other Names: Mizzou Nurse Workload and Well-Being Study

SUMMARY:
This observational study will evaluate the feasibility of linking nursing workload to burnout and physiological well-being among acute care nurses. Researchers will collect data from three sources: hospital workforce management software, wearable health devices (Oura Rings), and validated surveys. Fifty nurses from intensive care and medical-surgical units at a level one trauma center will participate. The study will also include interviews to better understand workplace stressors. Findings will help identify patterns that contribute to burnout and guide the development of future interventions to support nurse well-being and improve workforce retention.

ELIGIBILITY:
Inclusion Criteria:

* RN participants must be at least 18 years of age.
* Must be a credentialed registered nurse (RN) working fulltime (≥0.75 FTE) in the MUHC University Hospital on the surgical or cardiac ICUs, surgical specialties, or the cardiovascular unit.
* Must own a smart phone capable of supporting latest version of the Oura app with internet connectivity (Apple iOS15 and higher; Android 8.0 and higher with Google Play services) and Bluetooth 4.0.
* Ability to wear an Oura ring daily, 7 days/ week (at least 22 hours/day), and adhere to study procedures.
* Able to complete informed consenting procedures.

Exclusion Criteria:

* Known allergy or sensitivity to components of Oura ring.
* RNs working part-time or per diem
* Travel nurses
* Known allergies to the Oura ring
* Ring finger sizes incompatible with Oura Ring Gen 3 sizes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Registered nurses (RNs) working in intensive care and medical-surgical units at MU Health Care
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Acceptability | Enrollment
  Acceptability is evaluated based on the number of people who were approached to participate in the study compared to the number of people who agreed to participate. Reported as a percentage rate.
Data completion rate | Enrollment through 10 weeks
  Reported as percentage rate of complete data obtained at baseline, 5 weeks, and 10 weeks
Retention rate | Enrollment through 10 weeks
  Reported as a percentage rate reflecting the number of participants participating at study completion compared to the number of participants participating at study commencement.
Heart rate | Enrollment through 10 weeks
  Reported as a numerical value reflecting beats per minute.
Heart rate variability | Enrollment through 10 weeks
  Reported as a numerical value in (milliseconds)
Sleep duration | Enrollment through 10 weeks
  Reported as the total sleep time (hours and minutes)
Sleep score | Enrollment through 10 weeks
  Reported as a numerical value (index value) ranging from 0-100
Resilience score | Enrollment through 10 weeks
  Reported as a numerical score (composite index value) ranging from 0-100
Patient Acuity score | From enrollment through the end of 10 weeks
  The Oracle Health Workload Management Clairvia system operationalizes patient acuity in terms of the intensity of care provided by nursing staff and allows for the direct care time required per patient to be quantified. This allows capture of RNs' workload across the working shift, creating an individualized utilization value that can reported as a numerical value (score).

SECONDARY OUTCOMES:
The Perceived Stress Scale | Baseline, Week 5, Week 10
  The Perceived Stress Scale (PSS) (r = .93) is a 10-item survey measuring general perceived stress over the past 1 month. Scores range 0 to 40; ≥ 14 suggests at least moderate perceived stress.
The Professional Quality of Life Scale | Baseline
  The Professional Quality of Life Scale (ProQOL) is a 30-item measure of burnout, well-being, and occupational stress from the past 30 days. ProQOL subscales include compassion satisfaction (Cronbach's α = 0.88), burnout (Cronbach's α = 0.75), and secondary traumatic stress (Cronbach's α = 0.81). Scores are interpreted as ≤ 22 (low), 23-41 (moderate), and ≥42 (high) levels of the construct being measured.
The PROMIS-29 Profile v2.0 | Baseline, Week 5, Week 10
  The PROMIS®-29 Profile v.2.0 assesses 7 domains of mental and physical health, including anxiety, depression, fatigue, physical function, social role, sleep disturbance, pain. Raw scores are converted to T-scores with higher T-scores representing more of the construct being measured.
Feasibility of Intervention Measure (FIM) | Week 5, Week 10
  The Feasibility of Intervention Measure (FIM) is a 4-item, validated implementation outcome survey tool designed to assess how practical and achievable an intervention is within a given setting. Responses range from completely disagree to completely agree.
Acceptability of Intervention Measure (AIM) | Week 5, Week 10
  The AIM is a 4-item tool that evaluates the extent to which participants perceive an intervention as agreeable, satisfactory, or appealing. Responses range from completely disagree to completely agree.
Intervention Appropriateness Measure (IAM) | Week 5, Week 10
  The IAM is a 4-item tool that assesses the perceived fit or suitability of an intervention for a specific setting. Responses range from completely disagree to completely agree.
Qualitative Insights on Burnout and Organizational Stressors | Baseline
  Thematic analysis of semi-structured interviews exploring nurses' perceptions of stress, workload, and well-being.
Hours worked per week | Baseline through week 10
  Numerical value reflecting the total number of hours a nurse worked each week.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hulett, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot feasibility study involving sensitive biometric and survey data from a small sample of nurses. Individual participant data (IPD) will not be shared publicly due to privacy considerations and the exploratory nature of the study.